CLINICAL TRIAL: NCT02958436
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of Intravenously or Subcutaneously Administered REGN3500 in Healthy Adult Subjects
Brief Title: A Study of Intravenously or Subcutaneously Administered REGN3500 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R3500-HV-1551; 2016-002012-41 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-11-08 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Pharmacokinetics; REGN3500
MeSH Terms: interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Dose regimen 1 of REGN3500 (IV) versus placebo
  Interventions: Drug: REGN3500; Drug: Placebo
- Cohort 2 (Experimental): Dose regimen 2 of REGN3500 (IV) versus placebo
  Interventions: Drug: REGN3500; Drug: Placebo
- Cohort 3 (Experimental): Dose regimen 3 of REGN3500 (IV) versus placebo
  Interventions: Drug: REGN3500; Drug: Placebo
- Cohort 4 (Experimental): Dose regimen 4 of REGN3500 (SC) versus placebo
  Interventions: Drug: REGN3500; Drug: Placebo
- Cohort 5 (Experimental): Dose regimen 5 of REGN3500 (IV) versus placebo
  Interventions: Drug: REGN3500; Drug: Placebo

INTERVENTIONS:
Drug: REGN3500
Drug: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of single ascending intravenous (IV) and subcutaneous (SC) doses of REGN3500 in healthy adult males and females

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index</= 33 kg/m2
* In good health based on medical history, physical examination, vital signs, and laboratory testing
* Normal electrocardiogram (ECG) and blood pressure
* Able to comply with clinic visits and study-related procedures
* Able to sign an informed consent

Exclusion Criteria:

* Significant abnormalities in hematology, clinical chemistry, urinalysis, medical history
* Current smoker or recent history (within 3 months)
* History of tuberculosis, HIV, or hepatic disease
* Known sensitivity to doxycycline or other ingredients of study drug
* History of multiple/severe allergies
* Pregnant or breastfeeding women, or not currently using adequate contraception
* Participation in another investigational drug study within 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06-18 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events in subjects treated with REGN3500 | Up to 293 days after dosing

SECONDARY OUTCOMES:
Obtain the pharmacokinetic parameters (Cmax) that describe the serum concentration time profile of REGN3500 | Obtain serum samples pre-dose, immediately post-dose (infusion or injection end), 1, 2, 4, 8 (for subcutaneous) and 12 (for intravenous) hours after dosing
Obtain the pharmacokinetic parameters (Tmax) that describe the serum concentration time profile of REGN3500 | Obtain serum samples pre-dose, immediately post-dose (infusion or injection end), 1, 2, 4, 8 (for subcutaneous) and 12 (for intravenous) hours after dosing
Obtain the pharmacokinetic parameters (AUClast) that describe the serum concentration time profile of REGN3500 | Obtain serum samples pre-dose, immediately post-dose (infusion or injection end), 1, 2, 4, 8 (for subcutaneous) and 12 (for intravenous) hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Site 1, Ghent, Belgium

REFERENCES:
- [Derived] Kosloski MP, Kalliolias GD, Xu CR, Harel S, Lai CH, Zheng W, Davis JD, Kamal MA. Pharmacokinetics and pharmacodynamics of itepekimab in healthy adults and patients with asthma: Phase I first-in-human and first-in-patient trials. Clin Transl Sci. 2022 Feb;15(2):384-395. doi: 10.1111/cts.13157. Epub 2021 Sep 29. PMID 34523807